CLINICAL TRIAL: NCT04781231
Title: Impact of Music Added to the Usual Treatment on the Anxiety of Patients Undergoing Outpatient Cataract Surgery With Topical Anesthesia: Randomized Controlled Trial
Brief Title: Impact of Music Added to the Usual Treatment on the Anxiety of Patients Undergoing Outpatient Cataract Surgery With Topical Anesthesia
Acronym: MUSICAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study coordinator's decision
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LRU_2020_7
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cataract Surgery; Anxiety
Keywords: Cataract surgery; Anxiety; MusicCare; Music
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Masking Description: Participant in the group Usual care are unaware of the other groups, in order to avoir the Hawthorne effect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MusicCare® device (Experimental): The device consists of a headset and a touch pad. The patient can choose the style of music he prefers among 5. The 'U-shaped sequence' offered by MusicCare® is based on the principle of hypnoanalgesia. Musical induction is personalized according to the patient's preference. It will gradually lead to a hypnotic state of consciousness modified by variations in musical components such as rhythm, frequencies, orchestral formation and volume. A listening session lasts about 20 minutes.
  Interventions: Device: MusicCare® device
- Device with quiet recorded music (Active Comparator): An mp3 device with headphones will be given to the patient. Caregivers will launch a quiet 20-minute music playlist
  Interventions: Device: Device with quiet recorded music
- Usual management of anxiety (Other)
  Interventions: Other: Usual management of anxiety

INTERVENTIONS:
Device: MusicCare® device — The device consists of a headset and a touch pad. The patient can choose the style of music he prefers among 5. The 'U-shaped sequence' offered by MusicCare® is based on the principle of hypnoanalgesia. Musical induction is personalized according to the patient's preference. It will gradually lead to a hypnotic state of consciousness modified by variations in musical components such as rhythm, frequencies, orchestral formation and volume. A listening session lasts about 20 minutes.
  Arms: MusicCare® device
Device: Device with quiet recorded music — An mp3 device with headphones will be given to the patient. Caregivers will launch a quiet 20-minute music playlist
  Arms: Device with quiet recorded music
Other: Usual management of anxiety — No specific intervention
  Arms: Usual management of anxiety

SUMMARY:
Most patients treated for cataract surgery benefit from a short outpatient course with topical local anesthesia.

Having to undergo surgery, especially on the eye, without being asleep, can be stressful. Sometimes waiting in a waiting room with other patients can increase this stress. Patient anxiety may increase blood pressure potentially leading to the prescription of nicardipine to allow surgery to be performed. The patient's anxiety also increases the surgeon's stress, which can alter the conditions for performing the intervention and increase the risk of intraoperative complications.

Besides the administration of anxiolytics, nurses have few options for patients with anxiety. However, the treatment response time is not always appropriate and the patient's cooperation during the procedure can sometimes be impaired.

The effect of music on preoperative anxiety has been evaluated in several studies and has shown a significant decrease in anxiety before surgery.

MusicCare® is a "digital treatment" based on the principles of hypnoanalgesia which has been tested in the management of patients with various pathologies (depression, Alzheimer's disease, chronic pain, etc.) and has shown relative effectiveness. the absence of intervention on the pain and anxiety of patients.

In the context of cataract surgery with topical local anesthesia, we would like to assess the contribution of offering the MusicCare® listening device on patients' anxiety about absence

ELIGIBILITY:
Inclusion Criteria:

* First cataract surgery (first eye)
* Patient scheduled for short outpatient cataract surgery with topical anesthesia

Exclusion Criteria:

* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Self-assessed anxiety score between the 3 groups Description | baseline day, before entering the operating room
  Self-assessed anxiety score on a visual analogue scale (VAS) from 0 to 10 (0 means no anxiety and 10 the maximum anxiety imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Robin BARRAUD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschuld, Paris, France

IPD SHARING:
Plan to Share IPD: No